CLINICAL TRIAL: NCT03367520
Title: Helping Veterans With SMI "StayQuit" From Smoking After Inpatient Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Melanie Bennett, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00071331
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: StayQuit Intervention

STUDY DESIGN:
Intervention Model Description: This project has two phases. Phase 1: Develop StayQuit materials and train the study interventionist. Phase 2: Implement StayQuit with 10-20 Veterans who are hospitalized on the inpatient psychiatric unit at the Baltimore VA Medical Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- StayQuit (Experimental): StayQuit offers 3 meetings during hospitalization and up 13 telephone calls. StayQuit begins in the hospital with an assessment of motivation to remain quit after discharge and a brief intervention to develop discrepancy between values and behaviors and generate change talk. Participants are also encouraged to try nicotine replacement therapy during the hospitalization and after discharge. Telephone counseling is brief and focused on managing withdrawal from nicotine, coping with cravings, and supporting use of NRT. The investigators will work with hospital staff as needed to ensure that nicotine replacement therapy is offered to participants during the inpatient stay and prescribed at discharge.
  Interventions: Behavioral: StayQuit

INTERVENTIONS:
Behavioral: StayQuit — StayQuit offers 3 meetings during hospitalization and up 13 telephone calls. StayQuit begins in the hospital with an assessment of motivation to remain quit after discharge and a brief intervention to develop discrepancy between values and behaviors and generate change talk. Participants are also encouraged to try nicotine replacement therapy during the hospitalization and after discharge. Telephone counseling is brief and focused on managing withdrawal from nicotine, coping with cravings, and supporting use of NRT. The investigators will work with hospital staff as needed to ensure that nicotine replacement therapy is offered to participants during the inpatient stay and prescribed at discharge.

SUMMARY:
Given the high prevalence and great cost of smoking for individuals with serious mental illness, an effective smoking cessation intervention for this group of smokers that begins in the hospital and continues following discharge is needed. The investigators will develop and pilot test StayQuit, a multifaceted smoking cessation intervention for smokers with serious mental illness that begins in the hospital and continues for three months after discharge. StayQuit will provide a personalized and tailored experience for smokers with serious mental illness at different levels of motivation to remain abstinent. In the hospital, StayQuit will include a brief motivational intervention that will help smokers relate sustained smoking cessation to their values and preferences, shore up motivation to stay quit, and gain experience using nicotine replacement therapy. This will be followed by cessation-focused discharge planning to engage Veterans in continued smoking cessation services with StayQuit staff. After discharge, StayQuit will offer 13 weeks (spread out over 3 months) of smoking cessation telephone counseling. The investigators will examine the feasibility of StayQuit by collecting both quantitative data on attendance and qualitative data on participants' experiences.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving inpatient care at the Baltimore VAMC inpatient psychiatric unit
* 18 years of age or older
* Self-reported smoking of 5+ cigarettes a day prior to hospitalization

Exclusion Criteria:

* Documented history of severe neurological disorder
* Intellectual developmental disorder indicated by chart review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Attendance at in-person StayQuit sessions | 4 weeks
  Number of in-person StayQuit sessions a participant completes
Attendance at telephone StayQuit sessions | 13 weeks
  Number of telephone StayQuit sessions a participant completes

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No